CLINICAL TRIAL: NCT02072785
Title: Phase III Study of Vincristine Sulfate Liposome Or Vincristine Sulfate For Injection Combined Chemotherapy as Initial Induction Regimen In Adults Acute Lymphoblastic Leukemia
Brief Title: Phase III Study of Vincristine Sulfate Liposome For Injection In Adults With Naïve Acute Lymphoblastic Leukemia
Acronym: LY01609
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Luye Sike Pharmaceutical Co., Ltd. (Industry)
Collaborators: Ethics Committee of Blood Diseases Hospital (Unknown); Guangdong Provincial People's Hospital (Other); Qilu Hospital of Shandong University (Other); Xijing Hospital (Other); Xinqiao Hospital of Chongqing (Other); China Medical University, China (Other); West China Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Xuzhou Medical University (Other); First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUYESIKE-VSL-Ⅲ-01
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2013-11

CONDITIONS: Adult Acute Lymphoblastic Leukemia
Keywords: Adult Acute Lymphoblastic Leukemia; Vincristine Sulfate Liposome; Vincristine Sulfate
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vincristine Sulfate Liposome (Experimental): Vincristine Sulfate For Injection simulation agent 1.4mg/m2,(2mg, maximum dose), iv, d1, d8, d15, d22. Vincristine Sulfate Liposome For Injection: 1.4mg/m2, (2mg, maximum dose), iv, d1, d8, d15, d22.
  Duration between these two agents should be more than 2.5h, and saline should be avoided for flushing before Vincristine Sulfate Liposome For Injection.
  Interventions: Drug: Vincristine Sulfate Liposome
- Vincristine Sulfate (Active Comparator): Vincristine Sulfate For Injection 1.4mg/m2,(2mg, maximum dose), iv, d1, d8, d15, d22. Vincristine Sulfate Liposome For Injection simulation agent: 1.4mg/m2,(2mg, maximum dose), iv, d1, 8, 15, 22.
  Duration between these two agents should be more than 2.5h, and saline should not be used for flushing before Vincristine Sulfate Liposome For Injection simulation agent.
  Interventions: Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Vincristine Sulfate Liposome
  Arms: Vincristine Sulfate Liposome
Drug: Vincristine Sulfate
  Arms: Vincristine Sulfate

SUMMARY:
The purpose of this study is to determine whether vincristine sulfate liposome could reduce less peripheral neuropathy than vincristine sulfate,and be as effective as vincristine sulfate in adults with Naïve Acute Lymphoblastic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* De novo untreated ALL patients diagnosed by the bone marrow morphology, immunophenotype.
* 65 ≥ Age (years) ≥ 18 , male or female,
* ECOG Performance status of 0, 1, or 2.
* Patients must fulfill the following laboratory values

  1. Total bilirubin ≤2 ULN (corrected for same age)
  2. AST and ALT ≤3 ULN ( corrected for same ages)
  3. Serum creatinine ≤2 ULN (corrected for same age)
* Didn't receive any of the following treatments within 4 weeks before inclusion: chemotherapy, radiotherapy, replacement therapy, operation, long term of glucocorticoid therapy（>5 days）.
* No neurological disorders, no nerve or muscle injury (motor and sensory nerve).
* Patient must sign the informed consent and obey the protocol.

Exclusion Criteria:

* Atopy or allergic to multiple medicines or excipients.
* With serious complications that affect compliance.
* Serious organ dysfunctions or central nervous system disorders.
* Mixed phenotype acute leukemia, (T-B).
* Burkitt lymphoma/leukemia.
* Suspected or confirmed central nervous system leukemia.
* Diabetes.
* Received antifungal treatment with triazole agents within 1 month before inclusion.
* Reliance of antipyretic and analgesic medicines or psychotropic medicines.
* Undergoing or has undergone other clinical trials in 4 weeks before inclusion.
* Pregnant women, women of breast feeding or childbearing potential without contraception.
* Psychological disorders that affect signing consent.
* The investigators believe that patients who are not suitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(objectives (ORR) | up to 35 days
  ORR=CR+CRi CR(Complete response)
  1. No circulating blasts or extramedullary disease, No lymphadenopathy,splenomegaly,skin/gum infiltration/testicular mass/CNS involvement
  2. Trilineage hematopoiesis(TLH)and <5% blast in bone marrow
  3. ANC>1000/microl
  4. Platelets>100,000/microl
  CRi(Complete response with incomplete recovery of counts) Recovery of platelets but<100,000 or ANC is <1000/microl
Incidence of General peripheral neuropathy | A week before enrollment. one,two,three and four weeks after the start of induction chemotherapy
  Chemotherapy-induced peripheral neuropathy was evaluated By Total Neuropathy Score clinical Version(TNSc).
  If the score of any item of TNSc at anytime after the start of induction chemotherapy is higher than the baseline,it is considered that peripheral neuropathy occurs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Blood Diseases, Chinese Academy of Medical Sciences, Tianjin, China